CLINICAL TRIAL: NCT04065074
Title: A Single-arm, Open-label Study to Evaluate a Procedure for Intra-articular (IA) Injection of FX006 in Patients With Osteoarthritis (OA) of the Hip
Brief Title: Study to Evaluate a Procedure for Intra-articular Injection of FX006 in Patients With Osteoarthritis of the Hip
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FX006-2019-017
Record Dates: First submitted 2019-08-12; First posted 2019-08-22 (Actual); Results first posted 2020-12-01 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Osteoarthritis, Hip
Keywords: Osteoarthritis; Hip; Intra-articular; Injection
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis | interventions — FX006

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FX006 32 mg (Experimental): Single intra-articular (IA) injection of FX006 32 mg
  Interventions: Drug: FX006 32 mg

INTERVENTIONS:
Drug: FX006 32 mg — Extended-release 32 mg FX006 IA injection

SUMMARY:
This is a multi-center, single-arm, open-label study of FX006 in patients with hip OA. A maximum number of approximately 30 patients may be enrolled in this protocol. All enrolled patients will receive a single intra-articular (IA) injection of FX006.

DETAILED DESCRIPTION:
This is a multi-center, single-arm, open-label study in patients with hip OA to evaluate a procedure for intra-articular injection of FX006 in patients with hip OA. A maximum number of approximately 30 patients may be enrolled in this protocol.

All enrolled patients will receive a single intra-articular (IA) injection on Day 1 and be followed for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Willingness and ability to comply with the study procedures and visit schedules and ability to follow verbal and written instructions
* Patients 40 to 80 years of age, inclusive, on the day of consent
* Body Mass Index (BMI) ≤ 40 kg/m^2
* Has a documented clinical diagnosis of unilateral or bilateral hip OA for at least six months
* Kellgren-Lawrence (KL) Grade 2 or 3 in the index hip as confirmed by local read of X-ray obtained during Screening or ≤ 6 months of Screening visit
* Has clinically significant pain in the index hip

Exclusion Criteria:

* Has a history of hypersensitivity to triamcinolone acetonide, PLGA or lidocaine
* Is receiving anticoagulants (including warfarin, dabigatran, rivaroxaban, apixaban or low molecular weight heparin, ritonavir or cobicistat)
* Has had any previous surgery on the index hip
* Presence of surgical hardware or other foreign body in the index hip
* Has a history of infection of the index hip
* Has a diagnosis of other disorders in the index hip that can cause pain
* Has received any intra-articular injection in the index hip of corticosteroids, investigational (including FX006) or marketed (including Zilretta®) within the 3 months prior to Screening
* Has had trauma to the index hip in the past 3 months requiring immobilization
* Has a history or evidence of active or latent systemic fungal or mycobacterial infection (including tuberculosis), or of ocular herpes simplex
* Has within the past 3 months received corticosteroids by mouth, or by parenteral injection. Multiple courses or chronic intermittent use of inhaled, intranasal, or topical steroids is also exclusionary. Single courses of 14 days or less by those routes are permitted
* Has, at screening, or any time prior to day of scheduled injection (Day 1), clinical suspicion of local or systemic infection, including any infection in the index leg.
* Has a history of or active significant concomitant illness (known or suspected)
* Any bacterial or viral infection requiring parental antibiotics within 4 weeks of Day 1 or oral antibiotics within 2 weeks of Day 1
* Is a woman who is pregnant, nursing, lactating, or plans to become pregnant during the study
* Is a man who plans to conceive during the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2019-10-11 (Actual); Study Completion 2019-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Kelley, Study Director — Pacira Pharmaceuticals, Inc
Locations (5):
- United States (5):
  - Noble Clinical Research, Tucson, Arizona
  - Hope Clinical Research, Canoga Park, California
  - Biosolutions Clinical Research Center, La Mesa, California
  - Dream Team Clinical Research, Pomona, California
  - Lenox Hill Hospital, New York, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FX006 32 mg
Started | 16
Completed | 14
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Protocol Non-Compliance after injection | 1

BASELINE CHARACTERISTICS:
Arm/Group | FX006 32 mg
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (7.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.56 (6.785)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Successful Study Drug Administrations
Description: Successful study drug administration, defined as Injector reporting complete study drug administration.
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | FX006 32 mg
Number analyzed (Participants) | 16
Participants | 12
Statistical Analysis 1: Comparison: FX006 32 mg; Test type: Other — Proportion of Successful Administrations; Proportion of Successful Administrations = 0.75, 90% CI 2-sided [0.51 to 0.90]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from signing of informed consent to Last Visit.
Arm/Group | FX006 32 mg
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 1/16
Other Adverse Events (participants affected / at risk) | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FX006 32 mg (N=16)
Subchondrial Insufficiency Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Only 16 of the planned 30 patients were enrolled in this trial as the procedure for intra-articular injection of FX006 in patients with hip OA did not reduce the incidence of incomplete study drug administrations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-07-11): https://cdn.clinicaltrials.gov/large-docs/74/NCT04065074/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-18): https://cdn.clinicaltrials.gov/large-docs/74/NCT04065074/SAP_001.pdf